CLINICAL TRIAL: NCT04203069
Title: Multicenter, Controlled, Randomized, Open Label, Clinical Study to Assess the Efficacy of Auto-Adjustable MOBIDERM® Autofit NIGHT-time Compression Armsleeve in the Management of Upper Limb LYMphedema in Maintenance Phase: LYMphoNIGHT Study
Brief Title: Auto-Adjustable MOBIDERM® Autofit NIGHT-time Compression Armsleeve in the Upper Limb LYMphedema in Maintenance Phase
Acronym: LYMphoNIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Collaborators: International Clinical Trials Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC29; ANSM (Other: 2019-A02216-51)
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Lymphedema of Upper Arm
Keywords: Lymphedema of upper arm; Auto-Adjustable MOBIDERM® Autofit Armsleeve; Compression garments; Maintenance phase

STUDY DESIGN:
Intervention Model Description: Prospective open-label RIPH 2 study multicenter, controlled, randomized, with two parallel groups.
Who Masked: Outcomes Assessor
Masking Description: For the same patient, all measurements will be performed as far as possible by the same health professional who doesn't have the knowledge of the patient's group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group : Day-time compression sleeve (Placebo Comparator): Control group : Patients will wear the Day-time compression sleeve : THUASNE lymphatrex (± mitten) during 90 days.
  Interventions: Device: Control group : Day-time compression sleeve
- Day-time compression sleeve and Night-time MOBIDERM Autofit (Experimental): Intervention group : Patients will wear the Day-time compression sleeve : THUASNE lymphatrex (± mitten) + night-time Auto-Adjustable MOBIDERM® Autofit Armsleeve device with the possibility to wear an additional MOBIDERM® glove if a patient has a finger edema during 90 days.
  Interventions: Device: Intervention group : Day-time compression sleeve and Night-time MOBIDERM® Autofit

INTERVENTIONS:
Device: Control group : Day-time compression sleeve — In the control group, patients wear only day-time compression garment : lymphatrex during 3 months.
  The protocol will require 3 visits during the maintenance phase.
  Visit 1 at day 0 (until 5 days after the end of hospital): includes the inclusion visit with the reception of devices and some evaluations (clinical examination, lymphedema volume, questionnaires, ultrasound on a patients sub-group).
  Visit 2 at 30 days after the inclusion : includes some evaluations (clinical examination, lymphedema volume, questionnaires, ultrasound on a patients sub-group)
  Visite 3 at 90 days after the inclusion : includes some evaluations (clinical examination, lymphedema volume, questionnaires, ultrasound on a patients sub-group).
  Arms: Control group : Day-time compression sleeve
Device: Intervention group : Day-time compression sleeve and Night-time MOBIDERM® Autofit — In the intervention group, patients wear a day-time compression garment : lymphatrex and the night-time compression garment : MOBIDERM AUTOFIT during 3 months.
  The protocol will require 3 visits during the maintenance phase.
  Visit 1 at day 0 (until 5 days after the end of hospital): includes the inclusion visit with the reception of devices and some evaluations (clinical examination, lymphedema volume, questionnaires, ultrasound on a patients sub-group).
  Visit 2 at 30 days after the inclusion : includes some evaluations (clinical examination, lymphedema volume, questionnaires, ultrasound on a patients sub-group)
  Visite 3 at 90 days after the inclusion : includes some evaluations (clinical examination, lymphedema volume, questionnaires, ultrasound on a patients sub-group).
  Arms: Day-time compression sleeve and Night-time MOBIDERM Autofit

SUMMARY:
This study aims to assess Auto-Adjustable MOBIDERM® Autofit Armsleeve effect on upper limb volume excess after 3 months of maintenance phase treatment in patients with secondary upper limb lymphedema following breast cancer.

Half of the patient will wear a day-time and night time compression garment (MOBIDERM Autofit) for 3 months during the maintenance phase, while the other half will only wear day-time compression garment.

DETAILED DESCRIPTION:
The gold standard treatment to achieve volume reduction of lymphedema is based on a Decongestive Lymphedema Therapy (DLT).that consists in 2 consecutive phases: the initial intensive phase which aim is to obtain maximal reduction of lymphedema volume and a second, the maintenance phase which aim is to maintain the initial volumetric reduction achieved during phase 1 as long as possible. The second maintenance phase mostly based on patient self-management of his treatment, is not strictly codified, but includes compression therapy, nutritional recommendations, skin cares, physical exercises and manual lymphatic drainage.

24 hours compression using garments or bandages seems to be crucial for long term management of lymphedema.

Garment and bandages prescriptions for daily treatment are a common practice in the maintenance phase but are often unsuitable for night treatment, as bandages are effective when well applied but are highly dependent on the patients' skills, and garments, due to their nature, can be poorly tolerated leading to low adherence from patients to self-management care. In the end, there is an unmet medical need for night treatment during maintenance phase. .

In this context THUASNE developed a specific night-time garment, for lymphedema maintenance phase. It is a standard Auto-Adjustable Armsleeve using the MOBIDERM® technology.

MOBIDERM® AUTOFIT is a standard self-adjusting compressive MOBIDERM® sleeve, with mitten.

Several small rigid straps are placed throughout the product to facilitate the passage of the arm, to adapt the garment to the morphology of each patient and to tighten it.

A first pilot randomized controlled study demonstrated some benefit to use MOBIDERM Autofit during night-time as an adjuvant treatment to daily compressive garment.

The objective of this new study is to confirm, using a more robust methodology, the effect of Auto-Adjustable MOBIDERM® Autofit Armsleeve on maintenance phase treatment, worn during the night, within the period at risk for the so called rebound effect as reported in several observational studies.

ELIGIBILITY:
Inclusion Criteria:

* Women responding positively to the lymphedema reduction phase defined by a ≥ 20% decrease in lymphedema volume at the end of DLT
* Unilateral secondary upper limb lymphedema of stage II or III according to the criteria defined by the International Society of Lymphology, following breast cancer
* Affected arm that fits with one of the 6 standard sizes of the Auto-Adjustable MOBIDERM® Autofit armsleeve provided
* Signed informed consent prior to any study-mandated procedure
* Affiliated to the General regime of the Social Security or covered by a similar health insurance system

Non-inclusion criteria :

* Stage I lymphedema or located in several places
* Active cellulitis / Infectious dermo-hypodermatitis
* Lymphedema associated with active cancer needing acute chemotherapy
* Motor and sensitive neurological deficiency / psychiatric or addictive disorders
* Post-operative edema (i.e acute edema occurring during the days following breast cancer-related surgery)
* Patients for whom compression is contraindicated, such as untreated infections, skin irritation, thrombosis, presence of skin lesions on the armsleeve placement
* Pregnant or breastfeeding patient
* Previous history of hypersensitivity to MOBIDERM® technology or lymphatrex garment General conditions
* Participation to any other clinical study which has an impact on the different endpoints
* Unlikely to be followed up to 3 months with clinical assessment as per investigator's judgment
* Vulnerable patient according to the article L.1121-6 of the French Public Health Code, the adults being the object of a legal protective measure or enable to express their consent according to the article L.1121-8 of French Public Health Code

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
The volume excess variation | 90 days
  The primary endpoint of this study is to compare the volume excess variation of the upper limb between both groups from D0 to D90. Volume excess is defined as the volumetric difference between the affected upper limb compared to the contralateral upper limb, calculated with truncated cone formula.

SECONDARY OUTCOMES:
The quality of life (QoL): LYMQOL ARM self-questionnaire | 30 and 90 days
  The evolution of QoL is measured by LYMQOL ARM self-questionnaire and specific questions. This tool was designed as patient-completed questionnaire. The questions cover four domains : symptoms, body image/appearance, function, mood. Each item in each domain was scored : not at all (1), a little (2), Quite a bit (3), A lot (4). Specific questions are about patient's perception of benefit.
The range of motion | 30 and 90 days
  The evolution of range of motion of the arm is measured by joint movements : Antepulsion (flexion), retropulsion (extension), total abduction, adduction, lateral rotation (external rotation), medial rotation (internal rotation)
The volume excess variation | 30 days
  Volume excess is defined as the volumetric difference between the affected upper limb compared to the contralateral upper limb, calculated with truncated cone formula.
Patient's opinion on Global Impression of Change (PGI-C) | 30 and 90 days
  Patient's opinion on Global Impression of Change about her general condition is measured by the modified PGI-C questionnaire (Patient's opinion on Global Impression of Change). The scale has 7 levels from "no change or condition has got worsed"(worse outcome) to "a great deal better, and a considerable improvement that has made all the difference ( better outcome)". Intermediate levels are: "almost the same, hardly any change at all"; "a little better, but no noticeable change", "somewhat better, but the change has not made any real difference"; "moderately better, and a slight but noticeable change"; "better, and a definite improvement that has made a real and worthwhile difference.
Doctors' opinion on improving the patient's health condition (Clinical Global Improvement Impression) | 30 and 90 days
  Doctors' opinion on improving the patient's health condition caused by lymphedema is measured by the CGI-I modified questionnaire (Clinical Global Improvement Impression). This questionnaire allows doctors to evaluate the improvement of patients. The scale has 7 levels from "very strongly improved"(better outcome) to "very strongly aggravated"(worse outcome).Intermediate levels are: " Significantly improved " ; " Slightly improved " ; " No improvement " ; " Slightly aggravated " ; " Seriously aggravated ".
Doctors' opinion on severity about the lymphedema (CGI-S) | 30 and 90 days
  Doctors' opinion on severity about the lymphedema is measured by CGI-S. This questionnaire assesses the severity of lymphedema. This scale has 7 levels from "normal, not sick at all" (better outcome) to " among the most severely ill patients "(worse outcome). Intermediate levels are: " borderline ill " ; " slightly ill " ; " moderately ill " ; " clearly ill " ; " severely ill ".
number of days/nights : The compliance to treatment | 30 and 90 days
  The compliance to treatment (day-time and night-time only for Intervention Group) is reported by the physician in the e-CRF according to the patient diary. The compliance is measured in number of days and or nights (groupe I) when the device was worn and the average wearing time was : Full day/night, >50% of the day/night,<50% of the day/night
The evolution of quality of sleep: Jenkins self-questionnaire | 30 and 90 days
  The evolution of quality of sleep is measured by Jenkins self-questionnaire. This scale is composed of four questions about the quality of sleep.
The satisfaction about the device: questionnaire | 90 days
  Patient's satisfaction with regards to MOBIDERM® Autofit for patients from intervention group only by a satisfaction questionnaire. This questionnaire is focused on the product positioning and the comfort.
Number and type of serious and non-serious Adverse Device Effects | 90 days
  Number and type of serious and non-serious Adverse Device Effects (ADE) with a focus on cutaneous ADE will be reported during the study.
The elastometry | 30 and 90 days
  To compare the evolution of skin thickness, elasticity, suppleness on a subgroup of patients by ultrasound.
The percentage of patients presenting with a failure of maintenance | 30 and 90 days
  Percentage of patients presenting with a failure of maintenance phase, defined by a volume increase ≥ 30% of the volume reduction observed during intensive phase of decongestive lymphedema therapy (DLT)
The satisfaction about the daytime device: questionnaire | 90 days
  Patient's satisfaction with regards to daytime device for all patients by a satisfaction questionnaire. This questionnaire is focused on the product positioning and the comfort.
The quality of life (QoL): EQ-5D-5L self-questionnaire | 30 and 90 days
  The evolution of QoL is measured by EQ5D 5L self-questionnaire. This tool was designed as patient-completed questionnaire. The questions cover five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: ISABELLE QUERE, PUPH,MD, Principal Investigator — University Hospital, Montpellier
Locations (8):
- France (7):
  - Chu Grenoble, Grenoble
  - Chu Montpellier, Montpellier
  - Ghr Mulhouse, Mulhouse
  - CHU NICE, Nice
  - Nimes, Nîmes
  - Chu Toulouse, Toulouse
  - CHRU Tours, Tours
- Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quere I, Presles E, Coupe M, Vignes S, Vaillant L, Eveno D, Laporte S, Leizorovicz A; POLIT Study investigators. Prospective multicentre observational study of lymphedema therapy: POLIT study. J Mal Vasc. 2014 Jul;39(4):256-63. doi: 10.1016/j.jmv.2014.05.004. Epub 2014 Jun 12. PMID 24931830
- [Background] Mestre S, Calais C, Gaillard G, Nou M, Pasqualini M, Ben Amor C, Quere I. Interest of an auto-adjustable nighttime compression sleeve (MOBIDERM(R) Autofit) in maintenance phase of upper limb lymphedema: the MARILYN pilot RCT. Support Care Cancer. 2017 Aug;25(8):2455-2462. doi: 10.1007/s00520-017-3652-5. Epub 2017 Mar 9. PMID 28281052
- [Background] Brown JC, Cheville AL, Tchou JC, Harris SR, Schmitz KH. Prescription and adherence to lymphedema self-care modalities among women with breast cancer-related lymphedema. Support Care Cancer. 2014 Jan;22(1):135-43. doi: 10.1007/s00520-013-1962-9. Epub 2013 Sep 7. PMID 24013569